CLINICAL TRIAL: NCT02083809
Title: A Randomized Double-blinded Controlled Trial Comparing Dilation and Evacuation Outcomes With and Without Oxytocin Use
Brief Title: Effects of Oxytocin on Bleeding Outcomes During Dilation and Evacuation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Hawaii (Other)
Collaborators: Society of Family Planning (Other); University of Washington (Other)
Responsible Party: Principal Investigator, Bliss Kaneshiro, Professor of Obstetrics & Gynecology, University of Hawaii
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OxyDE
Record Dates: First submitted 2014-03-04; First posted 2014-03-11 (Estimated); Results first posted 2020-11-27 (Actual); Last update posted 2020-11-27 (Actual); Status verified 2020-11

CONDITIONS: Abortion; Dilation and Evacuation; Hemorrhage; Blood Loss
MeSH Terms: conditions — Dilatation, Pathologic; Hemorrhage | interventions — Electrolytes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): 500ml saline or lactated ringer without oxytocin added
  Interventions: Drug: Intravenous Fluids and Electrolytes
- Treatment group (Active Comparator): Intravenous oxytocin mixed with saline or lactated ringer
  Interventions: Drug: intravenous oxytocin

INTERVENTIONS:
Drug: intravenous oxytocin — 30 units of oxytocin added to 500ml of inert IV fluid (saline, lactated ringer)
  Arms: Treatment group
Drug: Intravenous Fluids and Electrolytes — 500 ml of inert IV fluid
  Arms: Placebo

SUMMARY:
Currently, there is very little research to identify ways to decrease blood loss during D&E (dilation and evacuation) procedures. The objective is to determine whether routine use of intravenous oxytocin will improve bleeding outcomes at the time of D&E at 18-24-weeks gestation. To evaluate the hypothesis, investigators will perform a randomized, double-blinded, placebo-controlled trial. The patient will be followed until discharged from the postoperative care unit during which time patient satisfaction, pain score and postoperative bleeding will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Requesting pregnancy termination
* Intrauterine pregnancy at 18- to 24-weeks gestation
* Gestational-age to be confirmed by ultrasound
* Patients with fetal anomaly or intrauterine fetal demise that occurred at 18- to 24-weeks gestation
* Willing and able to understand and sign written informed consents in English or Spanish and comply with study procedures

Exclusion Criteria:

* Ultrasound findings suggestive of placenta accreta
* Patients requiring preoperative misoprostol

Ages: 14 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 166 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-02 (Actual); Study Completion 2018-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Hawaii, Honolulu, Hawaii
  - University of Washington, Seattle, Washington

REFERENCES:
- [Derived] Whitehouse K, Tschann M, Soon R, Davis J, Micks E, Salcedo J, Savala M, Kaneshiro B. Effects of Prophylactic Oxytocin on Bleeding Outcomes in Women Undergoing Dilation and Evacuation: A Randomized Controlled Trial. Obstet Gynecol. 2019 Mar;133(3):484-491. doi: 10.1097/AOG.0000000000003104. PMID 30741801

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | Treatment Group
Started | 82 | 84
Completed | 78 | 82
Not Completed | 4 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Treatment Group | Total
Number analyzed (Participants) | 78 | 82 | 160
Age, Continuous [Mean (Standard Deviation); unit: age] | 27.2 (7.2) | 25.4 (7) | 26.3 (7.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 78 | 82 | 160
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 14 | 13 | 27
  Native Hawaiian or Other Pacific Islander | 23 | 27 | 50
  Black or African American | 5 | 10 | 15
  White | 36 | 32 | 68
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Rate at Which Providers Intervene to Control Blood Loss During D&E Procedures.
Time Frame: During surgical procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | Treatment Group
Number analyzed (Participants) | 78 | 82
Participants | 13 | 6

ADVERSE EVENTS:
Time Frame: 1 day
Description: laceration of the cervix requiring repair with suturing
Arm/Group | Placebo | Treatment Group
All-Cause Mortality (participants affected / at risk) | 0/78 | 0/82
Serious Adverse Events (participants affected / at risk) | 1/78 | 1/82
Other Adverse Events (participants affected / at risk) | 0/78 | 0/82
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=78) | Treatment Group (N=82)
cervical laceration (Reproductive system and breast disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT02083809/Prot_SAP_000.pdf